CLINICAL TRIAL: NCT06579261
Title: The Effects of Core Shamanism in Fibromyalgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Richard Edmund Harris, Samueli Endowed Chair and Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3326
Record Dates: First submitted 2024-08-06; First posted 2024-08-30 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-10

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia chronic pain
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fibromyalgia participants - Shamanic Intervention (Experimental)
  Interventions: Other: Core Shamanism

INTERVENTIONS:
Other: Core Shamanism — Each Shamanic intervention session, led by the shamanic practitioner, will include classical music as a control, followed by repetitive drumming and/or rattling music which the participant and shamanic practitioner will listen to for 15-30 mins. Following listening to drumming, the patient will then talk with the shamanic practitioner to debrief the experience of each session. Participants will also listen to classical music as a control stimulus.

SUMMARY:
This study aims to determine the feasibility of a shamanism intervention for patients with fibromyalgia, acquire efficacy data to determine if Shamanism reduces clinical pain and other common symptoms associated with fibromyalgia, and determine if the Shamanism intervention changes heart rate electrocardiogram (ECG), breathing rate, and brain wave electroencephalogram (EEG) outcomes in fibromyalgia patients and shamanic practitioners.

The investigators hypothesize that 80% of individuals will complete at least 80% of study visits, clinical pain severity and/or interference will be significantly reduced following the Shamanic intervention, and lung, heart, and/or brain activity will be altered with the Shamanic intervention and also become more synchronized between Shamanic Practitioners (SPs) and patients during the course of treatment.

DETAILED DESCRIPTION:
This study includes an 8-week long intervention, with 5 one-on-one treatment sessions with Fibromyalgia (FM) participants and shamanic practitioners (SPs). During each treatment session the FM participant will listen to classical music first as a control, followed by drumming music (4-7 beats/sec) for 15-30 minutes with the SP and a debrief session. The SP will employ the structure and principles of "Core Shamanism" as developed by Michael Harner. The first and last treatment sessions will include EEG measurements of both the patient and practitioner, while all sessions will have ECG and breathing rate for both patient and practitioner.

Pre screening questionnaires will be administered prior to shamanic treatments to ensure patients and SPs meet study inclusion criteria and give consent to the intervention. Following consent, pre and post treatment questionnaires will be administered to patient and SP participants to capture symptoms of fibromyalgia and treatment related experiences.

1-, 3-, and 6-month followup visits will involve the same questionnaires being administered and recorded to assess durability of treatment response.

ELIGIBILITY:
Inclusion Criteria for Fibromyalgia participants:

* Female
* Over 18 and under 75 years of age.
* Fibromyalgia patients and satisfies the 2016 Fibromyalgia Diagnostic Criteria for the classification of FM.
* Mean recalled pain over the last seven days (7-day recall) greater than or equal to 4 on a 10 cm Visual Analog Scale (VAS) for pain; 7-day recall.
* Willing to limit the introduction of any new medications or treatment modalities for control of FM symptoms during the study.
* Able to travel to the study site to receive shamanic treatments up to twice weekly.
* Understanding and willing to complete all study procedures.
* Capable of giving written informed consent.
* Proficient ability to speak, read, and write in english.

Exclusion Criteria:

* Presence of a concurrent autoimmune or inflammatory disease such as rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease, etc. that causes pain.
* History of head injury with substantial loss of consciousness
* Peripheral neuropathy of known cause that interferes with activities of daily living.
* Routine daily use of opioid analgesics, marijuana, or history of substance abuse.
* Stimulant medications, such as those used to treat Attention Deficit Disorder (ADD)/Attention-deficit/hyperactivity disorder (ADHD). (e.g., amphetamine/ dextroamphetamine [Adderall®], methylphenidate, dextroamphetamine), or the fatigue associated with sleep apnea or shift work (e.g., modafinil), are excluded.
* Concurrent participation in other therapeutic trials.
* Use of as needed (PRN) over the counter (OTC) pain medications (Nonsteroidal anti-inflammatory drugs (NSAIDs), etc.) on day of electroencephalogram (EEG) testing.
* Use of PRN opioid analgesics 48 hours prior to electroencephalogram (EEG) testing.
* Pregnant or nursing. A pregnancy test will be given prior to electroencephalogram (EEG) sessions.
* Severe psychiatric illnesses (current schizophrenia, major depression with suicidal ideation, substance abuse within two years).
* Contraindications to EEG methods. These may include but are not limited to: surgical clips, surgical staples, metal implants, and certain metallic dental material.
* Any impairment, activity or situation that is in the judgment of the Study Coordinator or Principal Investigator that would prevent satisfactory completion of the study protocol. This includes unreliable, or inconsistent pain scores as deemed by the principal investigator.
* Sufficient knowledge of Shamanism techniques that may bias participant outcomes.
* Presence of factors that may preclude the safe use of the Shamanism intervention.
* History vascular surgery in lower limbs or current lower limb vascular dysfunction.
* Presence of uncontrolled cardiovascular disease.
* Subjects with Worker's Compensation, Workman's Compensation, civil litigation or disability claims pertinent to the subject's fibromyalgia; current involvement in out-of-court settlements for claims pertinent to the subject's fibromyalgia; or currently receiving monetary compensation as a result of any of the above.
* Inability or unwillingness of an individual to give written informed consent.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study will only include women as most individuals with Fibromyalgia (FM) are female. Studying males is not optimal as a study including males would not have the required power with a large enough sample size. There are not enough males to be recruited in the study given the limited resources. This study will be powered well with a female population. Shamanic Practitioners (SPs) can be either male or female.
Enrollment: 25 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Primary Outcomes: Attendance Measurement | Pre screening (2-4 weeks prior to start of treatment visits), Baseline (Pre treatment visit Day 0), Treatment Visits 1-5 (To be done over 8 week long period), Post Treatment Assessment, 1-, 3-, and 6-month follow ups Post-treatment visit 5
  To investigate the primary outcome of feasibility, the investigators will record attendance and assess how many Fibromyalgia (FM) patients complete 80% of treatment visits (4 out of 5 sessions). Participants who complete at least 80% of visits will be marked as a completer and those who attend less than 80% of treatment visits will be marked as a "non-completer". The investigators will perform a completer versus non-completer analysis on all participants enrolled.

SECONDARY OUTCOMES:
Secondary Outcomes: Pain Measurement using Brief Pain Index (BPI) which uses a 0-10 numeric rating scale | Pre screening (2-4 weeks prior to start of treatment visits), Baseline (Pre treatment visit Day 0), Treatment Visits 1-5 (To be done over 8 week long period), Post Treatment Assessment, 1-, 3-, and 6-month follow ups Post-treatment visit 5
  Pain and other outcomes will be assessed at the University of California, Irvine by trained clinical research coordinators. The secondary outcomes for the study are pain severity and interference. These outcomes will be assessed with the Brief Pain Inventory (BPI). BPI is measured in the form of a participant self report questionnaire. It will measure where in the body pain is present and its severity as well as how much that pain is impacting daily life.
Secondary outcomes: Visual Analog Scale (VAS) Scales which uses a 10 cm visual scale. | Pre screening (2-4 weeks prior to start of treatment visits), Baseline (Pre treatment visit Day 0), Treatment Visits 1-5 (To be done over 8 week long period), Post Treatment Assessment, 1-, 3-, and 6-month follow ups Post-treatment visit 5
  Pain and other outcomes will be assessed at the University of California, Irvine by trained clinical research coordinators. The investigators will have each FM patient complete a 10 cm Visual Analog Scale (VAS) scale with anchors at 0 of "no pain" and 10 as "the worst pain imaginable". A VAS 7 day average recall will be used for inclusion into the study. Patients must score above a 4 on the VAS 7 day recall to be eligible to participate in this study. A daily VAS pain report and present VAS pain report will also be asked during screening, baseline, pre treatment, post treatment assessment visits, and 1-, 3-, and 6-month follow up visits.

OTHER OUTCOMES:
Exploratory Outcomes: Electrocardiogram (ECG) measured in millivolts and seconds or milliseconds (ms) | Treatment Visits 1-5 (To be done over 8 week long period)
  The investigators will collect ECG for all FM patients and Shamanic Practitioners (SPs) during all 5 treatment sessions. ECG will be performed using a Movesense sensor (commercially available) connected to a mobile device (via Bluetooth) which runs the patented electrocardio matrix (ECM) software. All data will be securely stored at University of California, Irvine.
Exploratory Outcomes: Electroencephalogram (EEG) measured in microvolts | Treatment Visits 1-5 (To be done over 8 week long period)
  The investigators will also collect EEG on patients and SPs during the first and last shamanic treatment session. The investigators will use the BrainVision EEG system to collect brain wave data from patients and SPs during the first and final treatment session. Two caps will be used, one for the patient and one for the SP, with both being attached to the EEG amplifier. All data will be securely stored at University of California, Irvine.
Exploratory Outcomes: Breathing Rate measured in breaths per minute | Treatment Visits 1-5 (To be done over 8 week long period)
  The investigators will collect breathing rates for all FM patients and SPs during all 5 treatment sessions. Breathing rate will be measured using a wearable device that does not interfere with the shamanic treatment sessions either. All data will be securely stored at University of California, Irvine.

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Richard, PhD, Principal Investigator — UCI SSIHI
Locations (1):
- Susan Samueli Integrative Health Institute, Irvine, California, United States